CLINICAL TRIAL: NCT02497872
Title: Early Precut Versus Pancreatic Duct Stent in Preventing Post-ERCP Pancreatitis in High-risk Subjects
Brief Title: Early Precut Versus Pancreatic Stent for Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Principal Investigator, Juan Lasa, MD, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERCP001
Record Dates: First submitted 2015-05-29; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Common Bile Duct Stones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Precut Sphincterectomy (Experimental): Biliary stone removal using early precut: Patients enrolled in this arm received biliary drainage through a small incision on the papilla with an endoscopic needle-knife - a technique called precut sphincterotomy.
  Interventions: Procedure: Biliary stone removal
- Pancreatic Duct Stent (Active Comparator): Biliary stone removal using persistence of cannulation and a later pancreatic duct stent placement: Patients enrolled in this arm received conventional biliary drainage through persistent biliary cannulation. After completion of biliary drainage, a prophylactic pancreatic duct stent was placed.
  Interventions: Procedure: Biliary stone removal

INTERVENTIONS:
Procedure: Biliary stone removal — Biliary stones are removed from the common bile duct by means of a sphincterotomy performed by standardized endoscopic retrograde cholangiopancreatography

SUMMARY:
BACKGROUND: The most common complication of endoscopic retrograde cholangiopancreatography (ERCP) is pancreatitis. Precut sphincterotomy has been regarded as a risk factor. However, early precut may actually reduce post-ERCP pancreatitis risk. However, early precut as a preventive measure has not been compared to other preventive measures, such as pancreatic duct stent placement.

AIM: To compare the efficacy of early precut sphincterotomy versus pancreatic duct stent placement in high-risk subjects undergoing ERCP.

MATERIALS AND METHODS: This is a single-blinded, randomized trial that took place in two tertiary referral centers in Buenos Aires. ERCP subjects shall present at least one of the following risk factors: female sex, age less than 40 years, clinical suspicion of Sphincter of Oddi dysfunction, previous pancreatitis, common bile duct diameter of less than 8 mm. Only those who present a difficult biliary cannulation shall be randomized into two groups: those who receive early precut sphincterotomy or those in whom persistency of biliary cannulation is intended with subsequent pancreatic duct stent placement after cholangiography is achieved. The incidence of post-ERCP pancreatitis as well as other complications shall be compared.

DETAILED DESCRIPTION:
It is well known that pancreatitis is the most common and dreadful complication of endoscopic retrograde cholangiopancreatography (ERCP). Historically, precut sphincterotomy has been regarded as a risk factor for post-ERCP pancreatitis. However, some evidence has suggested that if used at an early point during the procedure, it may actually behave as a protective factor.

In high risk patients, such as those patients with sphincter of Oddi dysfunction, pancreatic duct stent placement has been considered to be a prophylactic measure against pancreatitis. However, pancreatic duct stent placement can sometimes be a cumbersome procedure, and may require additional procedures (mainly if spontaneous stent dislodgment is not accomplished). There is no evidence comparing early precut versus pancreatic duct stent placement in high-risk patients.

As a consequence, the aim of this study was to compare the efficacy of early precut sphincterotomy versus pancreatic duct stent placement in patients presenting at least one risk factor for post-ERCP pancreatitis and difficult biliary cannulation.

A single-blinded, randomized trial was undertaken. Patients fulfilling inclusion criteria who presented with difficult biliary cannulation during ERCP were randomized to early precut or persistence in biliary cannulation with a sphincterotome with posterior pancreatic duct stent placement. The incidence of post-ERCP pancreatitis as well as other complications were compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with in need for ERCP due to benign or malignant biliopancreatic conditions, with at least one of the following features:
* female sex
* age less than 40 years
* clinical suspicion of Sphincter of Oddi Dysfunction
* previous pancreatitis
* common bile duct diameter of less than 8 mm
* Subjects with difficult biliary cannulation, as defined by previously published criteria

Exclusion Criteria:

* patients with contrast allergy
* pregnant women
* patients unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Post-ERCP Pancreatitis | 48 hours